CLINICAL TRIAL: NCT03252925
Title: A Safety and Efficacy Study of N-acetylcysteine in Patients With Transplant-Associated Thrombotic Microangiopathy
Brief Title: A Safety and Efficacy Study of NAC in Patients With TA-TMA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SOOCHOW-HY-2017
Record Dates: First submitted 2017-05-22; First posted 2017-08-17 (Actual); Results first posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2021-12

CONDITIONS: Thrombotic Microangiopathies; Hematologic Diseases
Keywords: N-acetylcysteine; Complement; Thrombotic Microangiopathies
MeSH Terms: conditions — Thrombotic Microangiopathies; Hematologic Diseases | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): N-Acetylcysteine
  Interventions: Drug: N-Acetylcysteine
- Control Group (Placebo Comparator): Placebo Oral Tablet
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: N-Acetylcysteine — 50mg/Kg.d, oral
  Other Names: NAC
  Arms: Experimental Group
Drug: Placebo Oral Tablet — 50mg/Kg.d, oral
  Other Names: Placebo
  Arms: Control Group

SUMMARY:
HSCT associated thrombotic microangiopathy(TA-TMA) is a heterogeneous, fatal disorder seen within 100 days post-transplant and presents with thrombocytopenia, hemolysis, acute renal failure, mental status changes and involvement of other organs. N-Acetylcysteine (NAC) is a small, simple molecule that began as a generic drug almost 40 years ago. It has since been approved by the FDA for many indications. The investigators conducted an prospective clinical trial to evaluate the safety and efficiency of NAC in patients with TA-TMA.

DETAILED DESCRIPTION:
Hematopoietic stem cell transplantation (HSCT) has been commonly used as a potentially curative option in the treatment of various hematological malignancies. However, it may end up with serious complications in various systems, including the hemostatic system. HSCT associated thrombotic microangiopathy(TA-TMA) is a heterogeneous, fatal disorder seen within 100 days post-transplant and presents with thrombocytopenia, hemolysis, acute renal failure, mental status changes and involvement of other organs. Since the pathophysiology has not been clarified, there are no established treatments for TA-TMA several agents seem to have successful results. N-Acetylcysteine (NAC) is a small, simple molecule that began as a generic drug almost 40 years ago. It has since been approved by the FDA for many indications. Studies showed NAC reduce plasma VWF multimers and VWF multimeric size without an effect on the bleeding time in vitro and in vivo, thus proposed as a possible supplementary treatment for TTP. The investigators conducted an prospective clinical trial to evaluate the safety and efficiency of NAC in patients with TA-TMA.

ELIGIBILITY:
Inclusion Criteria:

1. Patients be scheduled to undergo HSCT;
2. Not received decitabine 6 month ago;
3. Without severe organ damage;
4. ECOG 0-2;
5. Informed consent were obtained.

Exclusion Criteria:

1. Be sensitive to NAC;
2. Bronchial asthma；
3. Peptic ulcer；
4. Severe organ damage；
5. Pregnancy and breastfeeding women；

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Depei Wu, MD. PhD., Study Chair — The First Affiliated Hospital of Soochow University
Locations (1):
- The First affiliated Hospital of SooChow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] George JN, Lopez JA, Konkle BA. N-Acetylcysteine: an old drug, a new insight, a potentially effective treatment for thrombotic thrombocytopenic purpura. Transfusion. 2014 May;54(5):1205-7. doi: 10.1111/trf.12561. No abstract available. PMID 24819072
- [Background] Tersteeg C, Roodt J, Van Rensburg WJ, Dekimpe C, Vandeputte N, Pareyn I, Vandenbulcke A, Plaimauer B, Lamprecht S, Deckmyn H, Lopez JA, De Meyer SF, Vanhoorelbeke K. N-acetylcysteine in preclinical mouse and baboon models of thrombotic thrombocytopenic purpura. Blood. 2017 Feb 23;129(8):1030-1038. doi: 10.1182/blood-2016-09-738856. Epub 2016 Dec 23. PMID 28011677
- [Background] Acedillo RR, Govind M, Kashgary A, Clark WF. Treatment of severe, refractory and rapidly evolving thrombotic thrombocytopenic purpura. BMJ Case Rep. 2016 Jun 9;2016:bcr2016215491. doi: 10.1136/bcr-2016-215491. PMID 27284100
- [Background] Rottenstreich A, Hochberg-Klein S, Rund D, Kalish Y. The role of N-acetylcysteine in the treatment of thrombotic thrombocytopenic purpura. J Thromb Thrombolysis. 2016 May;41(4):678-83. doi: 10.1007/s11239-015-1259-6. PMID 26245827

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Group | Control Group
Started | 80 | 80
Completed | 66 | 74
Not Completed | 14 | 6
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 6 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- NAC Group: N-Acetylcysteine 50mg/Kg.d, oral
- Placebo Group: Placebo oral tablet 50mg/Kg.d, oral
- Total: Total of all reporting groups
Arm/Group | NAC Group | Placebo Group | Total
Number analyzed (Participants) | 66 | 74 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 11 | 18
  Between 18 and 65 years | 59 | 63 | 122
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 38 | 68
  Male | 36 | 36 | 72
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Yellow Race | 66 | 74 | 140
Region of Enrollment [Number; unit: participants]
  China | 66 | 74 | 140
Primary Diseases [Count of Participants; unit: Participants]
  Acute myeloid leukemia | 39 | 38 | 77
  Acute lymphoblastic leukemia | 15 | 18 | 33
  Aplastic anemia | 3 | 5 | 8
  Chronic myelogenous leukemia | 1 | 2 | 3
  Myelodysplastic syndrome | 7 | 10 | 17
  Lymphoma and multiple myeloma | 1 | 1 | 2
Transplant Type [Count of Participants; unit: Participants]
  HLA identical sibling | 14 | 16 | 30
  Related haplo-identical | 51 | 55 | 106
  Matched unrelated | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of TA-TMA.
Description: The incidence of TMA after HSCT.
Time Frame: 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | NAC Group | Placebo Group
Number analyzed (Participants) | 66 | 77
Participants | 5 | 15

2. Secondary Outcome: The Level of VWF Multimers
Description: The level of VWF multimers in patients post HSCT.
Time Frame: 100 days
Reporting Status: Not Posted

3. Secondary Outcome: The Level of Endothelial Micro Particle
Description: The level of endothelial micro particle in patients post HSCT.
Time Frame: 100 days
Reporting Status: Not Posted

4. Secondary Outcome: The Level of TNF-α
Description: The level of TNF-α in patients post HSCT.
Time Frame: 40 days
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | NAC Group | Placebo Group
Number analyzed (Participants) | 66 | 74
pg/mL | 0.4 [0 to 1.4] | 0.3 [0 to 2.1]

5. Secondary Outcome: The Level of ROS
Description: The level of ROS in patients post HSCT.
Time Frame: 100 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 100 days
Groups:
- Placebo: Placebo Oral Tablet 50mg/Kg.d, oral
Arm/Group | NAC Group | Placebo
All-Cause Mortality (participants affected / at risk) | 16/66 | 27/74
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/74
Other Adverse Events (participants affected / at risk) | 59/66 | 72/74
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NAC Group (N=66) | Placebo (N=74)
Abdominal pain or diarrhea (Gastrointestinal disorders) | 36 | 49
Hemorrhagic cystitis (Renal and urinary disorders) | 27 | 43
Fever (Blood and lymphatic system disorders) | 20 | 37
Upper gastrointestinal complications (Gastrointestinal disorders) | 3 | 18
Erythra (Blood and lymphatic system disorders) | 11 | 15
Cough or expectoration (Respiratory, thoracic and mediastinal disorders) | 9 | 15
Dizziness or headache (Vascular disorders) | 5 | 12
Gastrointestinal bleeding (Gastrointestinal disorders) | 6 | 6
Chest tightness (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Epilepsy (Nervous system disorders) | 1 | 4

LIMITATIONS AND CAVEATS:
Several outcome indicators are entirely inconsistent with our study's actual course of execution. First, the occurrence of TA-TMA was not limited to the first 100 days after hematopoietic stem cell transplantation. Secondly, the detection of VWF multimers, endothelial microparticles, and ROS was not performed according to the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT03252925/Prot_SAP_ICF_000.pdf